CLINICAL TRIAL: NCT01492439
Title: Examining the Effectiveness of Cognitive Remediation in a Supported Education Setting
Brief Title: Effectiveness of Cognitive Remediation in a Supported Education Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: George Brown College (Other)
Responsible Party: Principal Investigator, Sean Kidd, Principal Investigator, Independent Clinician Scientist and Head of Psychology Services, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 143/2011
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Psychosis
Keywords: Psychosis; Psychosis NOS; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Schizophrenia; Bipolar Disorder | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation and Supported Education (Experimental): Participants in this group will receive cognitive remediation training in addition to supported education. Cognitive remediation has two components: computer-based cognitive exercise sessions held on a twice weekly basis for 10 weeks as well as 10 weekly group discussion sessions (approximately 60 minutes in duration).
  Interventions: Behavioral: Cognitive Remediation
- Supported Education Only (Active Comparator): The George Brown College Redirection Through Education (RTE) is a supported education program, offered at no fee to students, that facilitates entry into formal education and employment for persons with mental illness (see http://www.georgebrown.ca/marketing/FTCal/access/C702.aspx for a full description). Participants in this arm will receive all services and supports provided by this program. However, they will not receive the additional cognitive remediation training provided to those randomized to the experimental arm of the study.
  Interventions: Behavioral: Supported Education

INTERVENTIONS:
Behavioral: Cognitive Remediation — The George Brown College Redirection Through Education (RTE) is a supported education program, offered at no fee to students, that facilitates entry into formal education and employment for persons with mental illness. In addition to the supports available to all RTE students, this group will receive a total of twenty 45 minute computer-based cognitive exercise sessions held twice a week using COGPACK (Ver 6.0,www.cogpack.de). This program facilitates practice across a range of cognitive functions, including attention,psychomotor speed,memory, and executive functions. Participants will also take part in 10 weekly group discussion sessions,approximately 60 minutes in duration, focusing on strategies for management of symptoms and other cognitive deficits in an academic setting.
  Other Names: CRT
  Arms: Cognitive Remediation and Supported Education
Behavioral: Supported Education — Students enroll in credit courses, such as communications, computer skills, and the psychology of human relations which can lead to eligibility for post-secondary programs. Remedial skills in English, supervised study skills classes and other non-credit courses are included. Vocational testing is offered to help students determine their interests and aptitudes and students try out possible careers as well as their readiness to return to work by engaging in volunteer and work placements. Counsellors are also available to assist students in areas such as learning difficulties and coping with the stresses of school. The overarching goal of this program is to help students explore valued non-illness identities, build confidence, and re-engage with their communities.
  Other Names: SE; RTE; Redirection Through Education
  Arms: Supported Education Only

SUMMARY:
The purpose of this study is to determine whether cognitive remediation as an adjunct to supported education, will result in improved cognitive functioning, symptoms, and performance in academic domains for persons with psychosis compared to supported education given alone.

DETAILED DESCRIPTION:
Cognitive remediation is an intervention that has been found effective in reducing the degree of the cognitive problems experienced by persons with schizophrenia. Investigators are proposing a project that will examine the effectiveness of cognitive remediation in a supported education setting at George Brown College in Toronto, Ontario. This study would build upon a feasibility study that the investigators have recently completed and represents an emerging line of inquiry as these interventions are increasingly being tested in community rehabilitation settings.

A large body of research has demonstrated the frequency of significant cognitive challenges among persons with schizophrenia who have ability levels that are, on average, 1-2 standard deviations lower than the general population in areas of problem solving, attention, and memory. These cognitive difficulties have been shown to have a marked impact on psychosocial functioning, making it very difficult to succeed for many people with schizophrenia in work and school settings. Work and school require people to prioritize, multi-task, sustain attention for prolonged periods, and remember material presented in a wide range of formats. Given the central role of education and employment in the recovery of persons with mental illness, it is crucial that efforts are made to address these cognitive difficulties to ensure the provision of a spectrum of services that can better address the quality of life of persons with schizophrenia.

In the past 10 years there has been a rapidly increasing interest in the development of means through which the impact of cognitive deficits might be ameliorated for persons with psychosis. This body of work has concentrated largely upon cognitive remediation strategies. Cognitive remediation (CR) refers to interventions in which a range of cognitive tasks are repeatedly practiced to improve attention, memory, and problem solving abilities. Most of these interventions are computer based, typically set up in the form of games, and others are paper-and-pencil.

Randomized controlled trials have consistently shown beneficial impacts of CR interventions on both cognitive and psychosocial functioning. Key findings include moderate effect sizes for improvements in attention, memory, and problem solving, more modest impacts on psychosocial functioning with better findings when CR is paired with supported employment. Less substantive impacts on psychosis symptomatology have been found, though self-esteem has been found to improve. Furthermore, the gains observed in CR have been found to be sustained for periods of up to 2 years post-intervention. Examination of non-specific effects has also indicated that CR leads to significant benefit over and above tasks that capture non-specific factors (e.g., computer skills training).

In general there has been a clear shift in the cognitive remediation literature towards examining functional outcomes and pairing cognitive remediation with other psychosocial interventions. This movement likely builds from criticisms of the narrow scope of earlier cognitive remediation studies which looked only at pre and post measures of cognitive functioning and their questionable association with 'real world' outcomes. In response to these criticisms Susan McGurk pioneered the examination of CR in supported employment contexts. To date, however, outside of the work of the present investigators, no studies of CR in supported education settings have been found. Research in this area is important because (1) education is a core component of the recoveries of people with severe mental illness and (2) cognitive impairments markedly limit what people might achieve in education settings.

Given the repeated calls in the literature for more randomized trials of cognitive remediation and the interest in the outcomes when partnered with psychosocial rehabilitation, this study addresses the following question: 'Does cognitive remediation as an adjunct to supported education result in improved cognitive functioning, symptoms, and performance in academic domains for persons with psychosis?'

This study will employ a randomized design in which term 1 students with psychosis will be randomized into either supported education alone (SE; n = 8) or supported education and cognitive remediation combined (SE + CR; n = 8).

The cognitive remediation intervention will have two components that will be completed over the course of 10 weeks within the academic term. First, participants will take part in a total of 20, 45 minute computer-based cognitive exercise sessions held on a twice weekly basis using COGPACK. This computer program facilitates practice across a broad range of cognitive functions, including attention and concentration, psychomotor speed, learning and memory, and executive functions. Participants will receive assistance on how to complete the cognitive exercises and will be given suggestions about strategies for improving performance on challenging exercises. In addition to computer exercises, participants will take part in 10 weekly group discussion sessions (approximately 60 minutes in duration). Topics in the group will include the role of cognitive factors in academic performance, the development of compensatory strategies for dealing with challenges in academic settings (e.g., study strategies, means of addressing attention difficulties), and strategies for managing difficulties such as anxiety and psychosis symptoms in school settings.

Evaluations will be completed at pre-intervention/control, post-intervention/control and 3 month follow up for both groups. The above sequence will be completed over the course of 5 academic terms to allow for a total sample of 64 (term 1 students are enrolled in every academic term and the 5th term would just be follow-up for the 4th group). Each trial within the academic term will be 10 weeks in length to allow for pre and post testing to take place within the term.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the George Brown Redirection Through Education program.
* A DSM-IV chart diagnosis of schizophrenia or other psychotic condition
* Stable use of medications for at least 3 months without plans of changing medications.
* Proficiency in English.

Exclusion Criteria:

* a psychiatric history of mental retardation, brain injury, or other neurological condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean A. Kidd, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - George Brown College, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Background] Anthony WA. Cognitive remediation and psychiatric rehabilitation. Psychiatr Rehabil J. 2008 Fall;32(2):87-8. doi: 10.2975/32.2.2008.87.88. No abstract available. PMID 18840561
- [Background] Bell M, Bryson G, Greig T, Corcoran C, Wexler BE. Neurocognitive enhancement therapy with work therapy: effects on neuropsychological test performance. Arch Gen Psychiatry. 2001 Aug;58(8):763-8. doi: 10.1001/archpsyc.58.8.763. PMID 11483142
- [Background] BERG EA. A simple objective technique for measuring flexibility in thinking. J Gen Psychol. 1948 Jul;39:15-22. doi: 10.1080/00221309.1948.9918159. No abstract available. PMID 18889466
- [Background] Davidson, L. (2003). Living Outside Mental Illness: Qualitative Studies of Recovery in Schizophrenia. New York City, NY: New York University Press.
- [Background] Delis, D., Kramer, J., Kaplan. E., & Ober, B. (1987). California Verbal Learning and Memory Test (Manual). San Antonio, TX: Psychological Corporation.
- [Background] Goeree R, Farahati F, Burke N, Blackhouse G, O'Reilly D, Pyne J, Tarride JE. The economic burden of schizophrenia in Canada in 2004. Curr Med Res Opin. 2005 Dec;21(12):2017-28. doi: 10.1185/030079905X75087. PMID 16368053
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] Health Canada. (2002). A Report on Mental Illnesses in Canada. Ottawa: Health Canada.
- [Background] Hodge MA, Siciliano D, Withey P, Moss B, Moore G, Judd G, Shores EA, Harris A. A randomized controlled trial of cognitive remediation in schizophrenia. Schizophr Bull. 2010 Mar;36(2):419-27. doi: 10.1093/schbul/sbn102. Epub 2008 Aug 20. PMID 18718884
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Kelland DZ, Lewis RF. The Digit Vigilance Test: reliability, validity, and sensitivity to diazepam. Arch Clin Neuropsychol. 1996;11(4):339-44. PMID 14588938
- [Background] Kurtz MM, Seltzer JC, Fujimoto M, Shagan DS, Wexler BE. Predictors of change in life skills in schizophrenia after cognitive remediation. Schizophr Res. 2009 Feb;107(2-3):267-74. doi: 10.1016/j.schres.2008.10.014. Epub 2008 Nov 8. PMID 19006657
- [Background] Kurtz MM, Seltzer JC, Shagan DS, Thime WR, Wexler BE. Computer-assisted cognitive remediation in schizophrenia: what is the active ingredient? Schizophr Res. 2007 Jan;89(1-3):251-60. doi: 10.1016/j.schres.2006.09.001. Epub 2006 Oct 27. PMID 17070671
- [Background] McGrew JH, Johannesen JK, Griss ME, Born DL, Katuin CH. Performance-based funding of supported employment for persons with severe mental illness: vocational rehabilitation and employment staff perspectives. J Behav Health Serv Res. 2007 Jan;34(1):1-16. doi: 10.1007/s11414-006-9045-z. Epub 2006 Dec 19. PMID 17180719
- [Background] Lezak, M. D. (1995). Neuropsychological Assessment. New York: Oxford University.
- [Background] Lindenmayer JP, McGurk SR, Mueser KT, Khan A, Wance D, Hoffman L, Wolfe R, Xie H. A randomized controlled trial of cognitive remediation among inpatients with persistent mental illness. Psychiatr Serv. 2008 Mar;59(3):241-7. doi: 10.1176/ps.2008.59.3.241. PMID 18308903
- [Background] McGurk SR, Mueser KT. Cognitive functioning, symptoms, and work in supported employment: a review and heuristic model. Schizophr Res. 2004 Oct 1;70(2-3):147-73. doi: 10.1016/j.schres.2004.01.009. PMID 15329293
- [Background] McGurk SR, Mueser KT, DeRosa TJ, Wolfe R. Work, recovery, and comorbidity in schizophrenia: a randomized controlled trial of cognitive remediation. Schizophr Bull. 2009 Mar;35(2):319-35. doi: 10.1093/schbul/sbn182. Epub 2009 Mar 5. PMID 19269925
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Medalia A, Richardson R. What predicts a good response to cognitive remediation interventions? Schizophr Bull. 2005 Oct;31(4):942-53. doi: 10.1093/schbul/sbi045. Epub 2005 Aug 24. PMID 16120830
- [Background] Mowbray CT, Bybee D, Collins ME. Follow-up client satisfaction in a supported education program. Psychiatr Rehabil J. 2001 Winter;24(3):237-47. doi: 10.1037/h0095088. PMID 11315210
- [Background] Radford LM, Chaney EF, O'Leary MR, O'Leary DE. Screening for cognitive impairment among inpatients. J Clin Psychiatry. 1978 Sep;39(9):712-5. PMID 690089
- [Background] Reeder C, Smedley N, Butt K, Bogner D, Wykes T. Cognitive predictors of social functioning improvements following cognitive remediation for schizophrenia. Schizophr Bull. 2006 Oct;32 Suppl 1(Suppl 1):S123-31. doi: 10.1093/schbul/sbl019. Epub 2006 Aug 10. PMID 16901950
- [Background] Rosenberg, M., (1965). Society and the Adolescent Self Image. Princeton, NJ: Princeton University Press.
- [Background] Reichenberg A, Harvey PD. Neuropsychological impairments in schizophrenia: Integration of performance-based and brain imaging findings. Psychol Bull. 2007 Sep;133(5):833-58. doi: 10.1037/0033-2909.133.5.833. PMID 17723032
- [Background] Rose, D., & Wykes, T., Farrier, D., Doran, A., Sporle, T., & Bogner, D. (2008). What do clients think of cognitive remediation therapy?: A consumer led investigation of satisfaction and side effects. American Journal of Psychiatric Rehabilitation, 11, 181-204.
- [Background] The Psychological Corporation. (1997). WAIS-III administration and scoring manual. San Antonio, TX: Psychological Corporation.
- [Background] Vauth R, Corrigan PW, Clauss M, Dietl M, Dreher-Rudolph M, Stieglitz RD, Vater R. Cognitive strategies versus self-management skills as adjunct to vocational rehabilitation. Schizophr Bull. 2005 Jan;31(1):55-66. doi: 10.1093/schbul/sbi013. Epub 2005 Feb 16. PMID 15888425
- [Background] Wilkinson ,G. (1993). Wide Range Achievement Test 3 (Manual). Wilmington, DE: Wide Range Inc.
- [Background] Wykes T, Huddy V. Cognitive remediation for schizophrenia: it is even more complicated. Curr Opin Psychiatry. 2009 Mar;22(2):161-7. doi: 10.1097/YCO.0b013e328322fbf4. PMID 19553870
- [Background] Wykes T, Reeder C, Williams C, Corner J, Rice C, Everitt B. Are the effects of cognitive remediation therapy (CRT) durable? Results from an exploratory trial in schizophrenia. Schizophr Res. 2003 Jun 1;61(2-3):163-74. doi: 10.1016/s0920-9964(02)00239-6. PMID 12729868

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Remediation + Supported Education: Participants in this group received cognitive remediation training in addition to supported education provided by the Redirection Through Education program at George Brown College. Cognitive remediation had two components: computer-based cognitive exercise sessions held twice a week for 10 weeks (approximately 45 minutes) and 10 weekly group discussion sessions (approximately 60 minutes).
- Supported Education Only: Participants in this group received all services and supports provided by the Redirection Through Education program at George Brown College. They did not receive the additional cognitive remediation training provided to those randomized to the experimental arm of the study.
Period: Overall Study
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Started | 19 | 18
Post-intervention | 18 | 13
Completed | 15 | 9
Not Completed | 4 | 9
Not completed — Withdrew from RTE | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Remediation + Supported Education: Participants in this group received cognitive remediation training in addition to supported education provided by the Redirection Through Education program at George Brown College. Cognitive remediation had two components: computer-based cognitive exercise sessions held twice a weekly for 10 weeks (approximately 45 minutes) and 10 weekly group discussion sessions (approximately 60 minutes).
- Total: Total of all reporting groups
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (12.3) | 34.7 (9.5) | 34.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Asian East | 1 | 2 | 3
  Asian South | 4 | 2 | 6
  Black Canadian | 2 | 1 | 3
  Black Caribbean | 2 | 1 | 3
  Mixed Background | 2 | 2 | 4
  White European Origin | 7 | 5 | 12
  Other | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 18 | 37
English as a second language [Number; unit: participants]
  Yes | 5 | 7 | 12
  No | 14 | 11 | 25
Self assessed level of competency in English [Number; unit: participants]
  Beginner | 2 | 0 | 2
  Intermediate | 9 | 15 | 24
  Advanced | 8 | 3 | 11
Primary diagnosis [Number; unit: participants]
  Schizophrenia | 11 | 10 | 21
  Schizoaffective | 1 | 2 | 3
  Bipolar | 5 | 2 | 7
  Psychosis NOS (Not otherwise specified) | 2 | 4 | 6
Hospitalized as a result of diagnosis [Number; unit: participants]
  Yes | 15 | 9 | 24
  No | 4 | 9 | 13
Housing [Number; unit: participants]
  Own/rent apartment or house | 5 | 6 | 11
  Supported housing e.g. boarding home | 3 | 4 | 7
  Live with family | 10 | 6 | 16
  Shelter or other temporary residence | 1 | 2 | 3
Years of education [Mean (Standard Deviation); unit: years] | 11.9 (1.2) | 13.2 (1.9) | 12.5 (1.7)
Years since diagnosis [Mean (Standard Deviation); unit: years] | 6.7 (6.5) | 7.0 (5.5) | 6.9 (5.9)
Years since last hospitalization [Mean (Standard Deviation); unit: years] | 3.2 (4.5) | 1.7 (2.9) | 2.5 (3.8)
Hours/week spent [Mean (Standard Deviation); unit: hours per week] — Meaningful activity is defined as time spent engaged in something meaningful that provides an individual with a sense of purpose.
  hours per week
    Competitive Employment | 1.7 (4.3) | 3.0 (6.9) | 2.4 (5.7)
    Student | 19.1 (1.5) | 19.7 (1.2) | 19.4 (1.3)
    Volunteer | 0.9 (2.1) | 1.7 (3.7) | 1.3 (3.0)
    Total hours engaged in meaningful activity | 21.8 (5.0) | 24.5 (7.1) | 23.1 (6.2)
Positive and Negative Syndrome Scale (PANSS) score [Mean (Standard Deviation); unit: units on a scale] — Symptoms of psychosis will be assessed using the Positive and Negative Syndrome Scale. The 30 item scale is comprised of 3 subscales measuring positive, negative and general psychopathology symptoms. Each item is scored using 7 anchoring criteria; 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores for the positive scale range from 7-49, the negative scale from 7-49, and general psychopathology 16-112, with total summed scores ranging from 30-210. 95>high, 75-95 medium and <75 low symptomology.
  units on a scale
    Positive | 13.58 (6.43) | 13.06 (3.95) | 13.32 (5.30)
    Negative | 13.42 (4.03) | 14.56 (4.95) | 13.97 (4.48)
    General psychopathology | 27.21 (6.87) | 28.33 (5.89) | 27.76 (6.35)
The Rosenberg Self-Esteem Scale Score [Mean (Standard Deviation); unit: units on a scale] — The Rosenberg Self Esteem Scale measures self esteem. This is a ten item, four point Likert scale with scores ranging from strongly agree to strongly disagree. Scores can range from 0-30. Total sum scores between 15 and 25 are within normal range; with scores below 15 suggest low self-esteem.
  units on a scale | 19.16 (4.63) | 17.39 (4.70) | 18.30 (4.69)
Performance on the California Verbal Learning Test [Mean (Standard Deviation); unit: Correct responses] — Verbal learning and memory will be assessed with the California Verbal Learning Test. A 9 word list is read to the participant (List A). Participants are asked to immediately free recall List A over 4 trials, then recall after a distractor task (short delay), then after a long delay.In the cued recall section, participants are asked to recall by category. In the long delay yes/no recognition, participants are asked to recall List A items out of a 27 word list. Higher repetitions and intrusions reveal greater impairment.
  Correct responses
    Trial 1 | 4.47 (1.35) | 4.50 (0.79) | 4.49 (1.10)
    Total free recall (trials 1-4) | 23.47 (4.13) | 23.50 (3.28) | 23.49 (3.69)
    Long delay free recall | 6.00 (1.70) | 5.61 (1.46) | 5.81 (1.58)
Performance on the Trail Making Test Part A [Mean (Standard Deviation); unit: Seconds] — The Trail Making Test Part A is a test involving using lines to connect numbers, it will be used to assess scanning ability and psychomotor speed. For this timed test, participants are scored by the number of seconds taken to complete the task, with high scores revealing greater impairment.
  Seconds | 49.00 (37.48) | 39.33 (15.96) | 44.30 (29.10)
Performance on the digit span subtest of the Wechsler Adult Intelligence Scale -III [Mean (Standard Deviation); unit: Correct responses] — Short term memory will be evaluated with the digit span subtest of the Wechsler Adult Intelligence Scale-III. Participants are asked to recall a sequence of numbers, starting with 2 and increasing to a sequence of 9 numbers. If the participant repeats the sequence correctly they score a one, if incorrect then score a zero. This test consists of two lists, one to be repeated forwards and the other backwards. The total score is a sum of sequences recalled correctly on the forward and backwards list.
  Correct responses
    Forward sequence | 9.58 (2.52) | 10.61 (2.30) | 10.08 (2.44)
    Backward sequence | 5.18 (2.22) | 6.17 (1.62) | 5.78 (1.97)
    Total | 14.74 (4.24) | 16.78 (3.08) | 15.73 (3.81)
Performance on the Trail Making Test Part B [Mean (Standard Deviation); unit: Seconds] — The Trail Making Test Part B assesses executive function. Trail Making Part B requires subjects to connect consecutively numbered and lettered circles by alternating between the 2 sequences. For this timed test, participants are scored by the number of seconds taken to complete the task, with high scores revealing greater impairment.
  Seconds | 98.68 (57.58) | 92.83 (42.93) | 95.84 (50.33)
Performance on the Wisconsin Card Sorting Test (WCST) [Mean (Standard Deviation); unit: Percentage of responses] — The WCST is a commonly used test of executive functioning that measures cognitive flexibility and problem solving skills. The 'number of categories' measures the number of correct responses. The percentage of perseverative errors provides the concentration of perseverative errors in relation to the overall test performance. The percentage conceptual level response provides the percentage of consecutive correct responses in runs of 3 or more.
  Percentage of responses
    % perseverative errors | 19.79 (12.23) | 18.94 (8.54) | 19.38 (10.46)
    % conceptual level of responses | 41.95 (26.20) | 52.94 (16.74) | 47.30 (22.51)
Performance on The Digit Vigilance Test [Mean (Standard Deviation); unit: Seconds] — The Digit Vigilance test measures sustained attention/vigilance. Participants are asked to cross out either 6s or 9s which appear randomly within 59 rows of 35 single digits. Scores are calculated for Total Time and Total Errors, with higher scores indicating greater impairment.
  Seconds | 458.37 (119.31) | 433.22 (103.34) | 446.14 (111.01)
Performance on The Digit Vigilance Test [Mean (Standard Deviation); unit: Incorrect responses] — The Digit Vigilance test measures sustained attention/vigilance. Participants are asked to cross out either 6s or 9s which appear randomly within 59 rows of 35 single digits. Scores are calculated for Total Time and Total Errors, with higher scores indicating greater impairment.
  Incorrect responses | 8.42 (6.59) | 6.72 (4.79) | 7.59 (5.77)
Performance on the Wisconsin Card Sorting Test [Mean (Standard Deviation); unit: Total categories] — The WCST is a commonly used test of executive functioning that measures cognitive flexibility and problem solving skills. The 'number of categories' measures the number of correct responses. The percentage of perseverative errors provides the concentration of perseverative errors in relation to the overall test performance. The percentage conceptual level response provides the percentage of consecutive correct responses in runs of 3 or more.
  Total categories | 36.37 (11.98) | 40.55 (7.82) | 38.41 (10.26)

OUTCOME MEASURES:

1. Primary Outcome: Completion of Academic Semesters
Description: During the study period, course instructors provided information as to whether participants had completed or withdrawn from academic semester 1 and 2. This data was used to determine whether completion of academic semesters might be explained by attending cognitive remediation alongside supported education. At the end of the each semester, course instructors notified the research team as to whether participants had completed or not completed the academic semester. The unit of measure, 'course completed' refers to the completion of the required number of courses in that academic semester to progress through to the next semester.
Time Frame: The end of the semester 1 (3 months following baseline) and semester 2 (6 months following baseline)
Measure: Mean (Standard Deviation); unit: Courses completed
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 19 | 18
Courses completed
  Semester 1 | 1.95 (0.29) | 1.67 (0.48)
  Semester 2 | 1.89 (0.375) | 1.67 (0.485)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.029, t-test, 1 sided — This applies to Semester 1
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.225, t-test, 1 sided — This applies to semester 2

2. Secondary Outcome: Positive and Negative Symptoms Scale (PANSS) Score at 3 Months
Description: Symptoms of psychosis will be assessed using the Positive and Negative Syndrome Scale. The 30 item scale is comprised of 3 subscales measuring positive, negative and general psychopathology symptoms. Each item is scored using 7 anchoring criteria; 1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme. Scores for the positive scale range from 7-49, the negative scale from 7-49, and general psychopathology 16-112, with total summed scores ranging from 30-210. 95>high, 75-95 medium and <75 low symptomology.
Time Frame: 3 months following baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
units on a scale
  Positive scale | 13.22 (5.32) | 13.90 (5.87)
  Negative scale | 12.83 (5.50) | 14.31 (4.25)
  General psychopathology scale | 27.89 (6.43) | 29.23 (7.81)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.247, ANCOVA — This applies to the 'positive' subscale of the PANSS
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.747, ANCOVA — This applies to the 'negative' subscale of the PANSS
Statistical Analysis 3: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.582, ANCOVA — This applies to the 'general psychopathology' subscale of the PANSS

3. Secondary Outcome: The Rosenberg Self-Esteem Scale Score at 3 Months
Description: The Rosenberg Self Esteem Scale measures self esteem. This is a ten item, four point Likert scale with scores ranging from strongly agree to strongly disagree. Scores can range from 0-30. Total sum scores between 15 and 25 are within normal range; with scores below 15 suggest low self-esteem.
Time Frame: 3 months following Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
units on a scale | 21.72 (3.75) | 15.31 (3.97)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.000, ANCOVA

4. Secondary Outcome: The Positive and Negative Symptoms Scale (PANSS) Score at 6 Months
Description: as for outcome 2
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
units on a scale
  Positive scale | 14.40 (6.27) | 13.44 (5.64)
  Negative scale | 11.53 (2.13) | 17.44 (6.02)
  General psychopathology scale | 26.20 (6.68) | 28.44 (7.62)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.950, ANCOVA — This applies to the 'positive' subscale of the PANSS
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.027, ANCOVA — This applies to the 'negative' subscale of the PANSS
Statistical Analysis 3: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.639, ANCOVA — This applies to the 'general psychopathology' subscale of the PANSS

5. Secondary Outcome: The Rosenberg Self-Esteem Scale Score at 6 Months
Description: as for outcome 3
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
units on a scale | 21.53 (4.31) | 16.00 (4.95)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.008, ANCOVA

6. Secondary Outcome: The California Verbal Learning Test at 3 Months
Description: Verbal learning and memory will be assessed with the California Verbal Learning Test. A 9 word list is read to the participant (List A). Participants are asked to immediately free recall List A over 4 trials, then recall after a distractor task (short delay), then after a long delay.In the cued recall section, participants are asked to recall by category. In the long delay yes/no recognition, participants are asked to recall List A items out of a 27 word list. Higher repetitions and intrusions reveal greater impairment.
Time Frame: 3 months following Baseline Assessment
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Correct responses
  Trial 1 | 5.83 (1.42) | 5.23 (1.54)
  Total free recall (Trials 1-4) | 28.28 (4.20) | 26.08 (4.03)
  Long delay free recall | 7.22 (1.26) | 6.92 (1.12)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.314, ANCOVA — This applies to Trial 1 on the CVLT
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.242, ANCOVA — This applies to the total score of trials 1-4 (total free recall) of the CVLT
Statistical Analysis 3: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.669, ANCOVA — This applies to the 'long delay free recall' subtest of the CVLT

7. Secondary Outcome: The California Verbal Learning Test at 6 Months
Description: as for outcome 6
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Correct responses
  Trial 1 | 6.00 (1.69) | 5.00 (1.12)
  Total free recall (Trials 1-4) | 28.60 (4.60) | 26.44 (2.40)
  Long delay free recall | 7.40 (1.64) | 7.44 (0.53)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.139, ANCOVA — This applies to the 'trial 1' subtest of the CVLT
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.269, ANCOVA — This applies to the total of trials 1-4 (total free recall) of the CVLT
Statistical Analysis 3: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.666, ANCOVA — This applies to the 'long delay free recall' subtest of the CVLT

8. Secondary Outcome: The Trail Making Test Part A at 3 Months
Description: The Trail Making Test Part A is a test involving using lines to connect numbers, it will be used to assess scanning ability and psychomotor speed. For this timed test, participants are scored by the number of seconds taken to complete the task, with high scores revealing greater impairment.
Time Frame: 3 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Seconds | 33.89 (16.73) | 27.08 (6.71)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.391, ANCOVA

9. Secondary Outcome: The Trail Making Test Part A at 6 Months
Description: as for outcome 8
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Seconds | 33.20 (16.21) | 31.00 (8.25)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.958, ANCOVA

10. Secondary Outcome: The Digit Span Subtest of the Wechsler Adult Intelligence Scale - III at 3 Months
Description: Short term memory will be evaluated with the digit span subtest of the Wechsler Adult Intelligence Scale-III. Participants are asked to recall a sequence of numbers, starting with 2 and increasing to a sequence of 9 numbers. If the participant repeats the sequence correctly they score a one, if incorrect then score a zero. There are two lists, one to be repeated forwards and the other backwards. The total score is a sum of sequences recalled correctly.
Time Frame: 3 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Correct responses
  Forward | 9.05 (2.09) | 9.07 (1.32)
  Backward | 5.22 (2.20) | 5.23 (1.36)
  Total | 14.28 (3.75) | 14.31 (1.89)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.754, ANCOVA — This applies to the 'forward' sequence of the Digit Span Test
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.518, ANCOVA — This applies to the 'backward' sequence of the Digit Span Test
Statistical Analysis 3: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.531, ANCOVA — This applies to the total score (forward+backwards) on the Digit Span Test

11. Secondary Outcome: The Digit Span Subtest of the Wechsler Adult Intelligence Scale - III at 6 Months
Description: as for outcome 10
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Correct responses
  Forward | 9.73 (2.25) | 9.67 (2.45)
  Backward | 6.60 (2.50) | 5.78 (1.99)
  Total | 16.33 (4.32) | 15.22 (4.18)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.802, ANCOVA — This applies to the 'forward' sequence of the Digit Span Test
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.091, ANCOVA — This applies to the 'backwards' sequence of the Digit Span Test
Statistical Analysis 3: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.171, ANCOVA — This applies to the total score (forward + backwards) on the Digit Span Test

12. Secondary Outcome: The Trail Making Test Part B at 3 Months
Description: The Trail Making Test Part B assesses executive function. Trail Making Part B is similar to Part A but is a more challenging task because it requires subjects to connect consecutively numbered and lettered circles by alternating between the 2 sequences. For this timed test, participants are scored by the number of seconds taken to complete the task, with high scores revealing greater impairment.
Time Frame: 3 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Seconds | 104.11 (73.32) | 81.31 (27.96)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.267, ANCOVA

13. Secondary Outcome: The Trail Making Part B at 6 Months
Description: as for outcome 12
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Seconds | 88.58 (66.98) | 70.22 (24.63)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.527, ANCOVA

14. Secondary Outcome: The Wisconsin Card Sorting Test at 3 Months
Description: The WCST is a commonly used test of executive functioning that measures cognitive flexibility and problem solving skills. The 'number of categories' measures the number of correct responses. The percentage of perseverative errors provides the concentration of perseverative errors in relation to the overall test performance. The percentage conceptual level response provides the percentage of consecutive correct responses in runs of 3 or more.
Time Frame: 3 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Percentage of responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Percentage of responses
  % perseverative errors | 19.56 (16.39) | 14.85 (8.93)
  % conceptual level of responses | 50.67 (26.61) | 60.31 (22.24)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.852, ANCOVA — This applies to the percentage of perseverative errors on the WCST
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.637, ANCOVA — This applies to the percentage of conceptual level responses on the WCST

15. Secondary Outcome: The Wisconsin Card Sorting Test at 3 Months
Description: The Wcst is a commonly used test of executive functioning that measures cognitive flexibility and problem solving skills. The 'number of categories' measures the number of correct responses. The percentage of perseverative errors provides the concentration of perseverative errors in relation to overall test performance. The percentage conceptual level response provides the percentage of consecutive correct responses in runs of 3 or more.
Time Frame: 3 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Correct responses | 40.00 (13.32) | 44.38 (9.39)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.612, ANCOVA — This applies to the total number of correct categories on the WCST

16. Secondary Outcome: The Wisconsin Card Sorting Task at 6 Months
Description: as for outcome 14
Time Frame: 6 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Percentage of responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Percentage of responses
  % perseverative errors | 21.27 (14.32) | 16.00 (10.39)
  % conceptual level of responses | 49.67 (26.18) | 53.78 (33.04)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.156, ANCOVA — This applies to the percentage of perseverative errors on the WCST
Statistical Analysis 2: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.926, ANCOVA — This applies to the percentage of conceptual level responses on the WCST

17. Secondary Outcome: The Wisconsin Card Sorting Task at 6 Months
Description: as for outcome 15
Time Frame: 6 months following baseline assessment
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Correct responses | 39.87 (12.36) | 41.33 (15.12)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; This applies to the total number of categories on the WCST; Test type: Superiority or Other; p = 0.843, ANCOVA

18. Secondary Outcome: The Digit Vigilance Test at 3 Months
Description: The Digit Vigilance test measures sustained attention/vigilance. Participants are asked to cross out either 6s or 9s which appear randomly within 59 rows of 35 single digits. Scores are calculated for Total Time and Total Errors, with higher scores indicating greater impairment.
Time Frame: 3 months following Baseline assessment
Measure: Mean (Standard Deviation); unit: Incorrect Responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Incorrect Responses | 8.33 (8.70) | 10.54 (8.67)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.129, ANCOVA — This applies to the total number of errors made on the DVT

19. Secondary Outcome: The Digit Vigilance Test at 3 Months
Description: as for outcome 18
Time Frame: 3 months following baseline assessment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 18 | 13
Seconds | 446.11 (111.97) | 366.61 (43.58)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; This applies to the total time taken to complete the DVT; Test type: Superiority or Other; p = 0.004, ANCOVA

20. Secondary Outcome: The Digit Vigilance Test at 6 Months
Description: as for outcome 18
Time Frame: 6 months following baseline assessment
Measure: Mean (Standard Deviation); unit: Incorrect Responses
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Incorrect Responses | 5.60 (3.70) | 5.22 (5.07)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; Test type: Superiority or Other; p = 0.853, ANCOVA; This applies to the total number of errors on the DVT

21. Secondary Outcome: The Digit Vigilance Test at 6 Months
Description: as for outcome 18
Time Frame: 6 months following baseline assessment
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Number analyzed (Participants) | 15 | 9
Seconds | 409.93 (89.16) | 433.33 (74.2)
Statistical Analysis 1: Comparison: Cognitive Remediation + Supported Education vs Supported Education Only; This applies to the total time taken to complete the DVT; Test type: Superiority or Other; p = 0.468, ANCOVA

ADVERSE EVENTS:
Time Frame: December 2011 - July 2013
Arm/Group | Cognitive Remediation + Supported Education | Supported Education Only
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No